CLINICAL TRIAL: NCT03551184
Title: Inflammation Och hjärnfunktion - Huvudstudie
Brief Title: Inflammation and Brain Function - Main Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: University of California, San Francisco (Other); The Swedish Society of Medicine (Other); Swedish Heart Lung Foundation (Other); The Swedish Research Council (Other Government); Swedish Council for Working Life and Social Research (Other); Stockholm University (Other)
Responsible Party: Principal Investigator, Mats Lekander, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: 2010/1363-32
Record Dates: First submitted 2018-05-29; First posted 2018-06-11 (Actual); Last update posted 2018-06-11 (Actual); Status verified 2018-05

CONDITIONS: Sickness Behavior
Keywords: Sickness behavior; Endotoxin; Lipopolysaccharide; Psychoneuroimmunology
MeSH Terms: conditions — Illness Behavior | interventions — Endotoxins; Lipopolysaccharides

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Endotoxin (Active Comparator): Endotoxin 0.6 ng/kg body weight injection
  Interventions: Biological: Endotoxin
- Placebo (Placebo Comparator): Saline injection
  Interventions: Biological: Placebo

INTERVENTIONS:
Biological: Endotoxin — Endotoxin at 0.6 ng/kg of body weight administered intravenously (Escherichia Coli, Lot nr G3E0609, United States Pharmacopeia Rockville, MD)
  Other Names: LPS; Lipopolysaccharide
  Arms: Endotoxin
Biological: Placebo — Saline administered intravenously
  Arms: Placebo

SUMMARY:
In this randomized double blind study, 52 healthy participants were injected with either 0.6 ng/kg body weight or placebo to test if changes in pain sensitivity is associated with change in neural activity using BOLD MR scanning.

DETAILED DESCRIPTION:
52 healthy participants were included in this randomized double blind study. Participants were injected once, and randomized to injection with with the active component or placebo. Participants were recruited by advertising and screened through questionnaires and a health examination by a physician. They were asked not to engage in strenuous physical activities, sleep regular hours and refrain from alcohol the day before the experiment. If the participants felt ill, e.g. coming down with a cold, they were instructed to call and were rescheduled for a later appointment. C-reactive protein (CRP) was assessed to exclude participants having an ongoing infection on the experimental day. Pregnancy was also an exclusion criteria and a pregnancy test was administered for all female participants on arrival. Pain sensitivity measures were tested at baseline and at peak inflammatory response 1-2 hours after injection. Both deep and cutaneous pain at threshold and suprathreshold noxious levels were tested. Heat- and cold (cutaneous) pain sensitivity was assessed for threshold stimuli and intense noxious stimuli, as well as pressure (deep) pain thresholds and CPM (descending pain inhibition). These tests were conducted while the participants were in the MR-scanner to investigate neural correlates to change in pain sensitivity. Subjects filled out questionnaires at baseline, 90 minutes, 3.5 and 5 hours after injection.

The study and the procedures used in the study are described in detail here: https://openarchive.ki.se/xmlui/bitstream/handle/10616/44650/Thesis_Bianka_Karshikoff.pdf?sequence=8&isAllowed=y

The following papers using data from this study is published:

Lindstedt F, Karshikoff B, Schalling M, Olgart Hoglund C, Ingvar M, Lekander M & Kosek E. Serotonin-1A Receptor Polymorphism (rs6295) Associated with Thermal Pain Perception. PLOS ONE. 2012;7(8):e43221. Epub 2012/09/07.

Karshikoff B, Jensen KB, Kosek E, Kalpouzos G, Soop A, Ingvar M, Olgart Höglund C, Lekander M, Axelsson J. Why sickness hurts: A central mechanism for pain induced by peripheral inflammation. Brain, Behavior, and Immunity 2016 Oct;57:38-46.

Lekander M, Karshikoff B, Johansson E, Soop A, Fransson P, Lundström J N, Andreasson A, Ingvar M, Petrovic P, Axelsson J/Nilsonne G. Intrinsic functional connectivity of insular cortex and symptoms of sickness during acute experimental inflammation. Brain, Behavior, and Immunity 2016 Aug;56:34-41.

Andreasson A, Wicksell RK, Lodin K, Karshikoff B, Axelsson J, Lekander M. A Global Measure of Sickness Behavior: Development of the Sickness Questionnaire (SicknessQ). Journal of Health Psychology. 2016 Jul 24.

Karshikoff B, Lekander M, Soop A, Lindstedt F, Ingvar M Kosek E, Olgart Höglund C, & Axelsson J. Modality and sex differences in pain sensitivity during human endotoxemia. Brain, Behavior, and Immunity. 2015 May;46:35-43

ELIGIBILITY:
Inclusion Criteria:

* Healthy subjects

Exclusion Criteria:

* Diagnosed physiological or psychiatric disease
* Needle anxiety or blood phobia
* Regular medication (excluding contraceptive pill)
* Infection in the last two weeks
* Pregnancy or breastfeeding
* Smoking
* Excessive alcohol use
* Body mass index in the range of obesity (>30 kg/m2) or underweight (<18.5 kg/m2)
* Invisible veins in the antecubital area of the arms
* Known or risk of metal inserted in body
* Claustrophobic tendensies

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 52 (Actual)
Dates: Start 2010-10 (Actual); Primary Completion 2011-03 (Actual); Study Completion 2011-03 (Actual)

PRIMARY OUTCOMES:
Pain sensitivity (cutaneous and deep) | 7.5 hours
  Both deep and cutaneous pain at threshold and suprathreshold noxious levels. Heat- and cold (cutaneous) pain sensitivity was assessed for threshold stimuli and intense noxious stimuli, as well as pressure (deep) pain thresholds and CPM (descending pain inhibition).
Brain function | 7.5 hours
  BOLD activity from MR scans
  1. Functional connectivity of the insular cortex during acute inflammation, in relation to symptoms of sickness.
  2. Changes in central pain mechanism during acute inflammation, assessed as activity in the insula and areas of the descending pain inhibitory pathways in the brain.
  3. Changes in brain function during an emotional task with an interoceptive component during acute inflammation.

SECONDARY OUTCOMES:
Self-rated health | 4.5 hours
  "How is your health right now?" rated on a 7 point Likert scale at baseline, after 90 minutes and after 4.5 hours.
  "How do you rate your general state of health?" rated on a 5-point Likert scale at 90 minutes post-injection
Facial appearence | 2 h
  Photos were taken under standardised conditions before and after injection

IPD SHARING:
Plan to Share IPD: Undecided